A Single Center, Randomized and Controlled Clinical Study of Inverted Internal Limiting Membrane Insertion Combined with Air Tamponade in the Treatment of Macular Hole Retinal Detachment in High Myopia

**Study Protocol** 

Version number: 2.0

Version date: April 2, 2017

Principal Investigator: Fenghua Wang

Department of Ophthalmology

Shanghai General Hospital

Version number: Version 2

### **Summary**

## 1. Purpose

To evaluate the surgical outcomes of inverted internal limiting membrane insertion combined with air tamponade in the treatment of macular hole retinal detachment (MHRD) in high myopia, and also to compare the treatment efficacy between different surgical approaches of MHRD.

## 2. Design

Design: a prospective, single-centered, randomized, controlled clinical trial

### 3. Target

Patients with high myopia complicated by macular hole associated-retinal detachment.

### 4. Inclusion Criteria

#### Inclusion Criteria

- 1) Prior written informed consent should be obtained before any assessment is carried out;
- 2) Participants are more than 18 years of age, and less than 75 years of age, male or female Chinese patients;
- Visual impairment is caused by macular hole associated with retinal detachment secondary to high myopia;
- 4) Axial length  $\geq$  26mm, or the refractive error  $\geq$  -6.0D

### 5. Exclusion criteria

## **Exclusion Criteria**

- 1) Failure to comply with research or follow-up procedures;
- 2) Diabetes with uncontrolled blood glucose (defined as fasting plasma glucose more than 7.0mmol/L or blood glucose more than 11.1mmol/L 2 hours postprandial), and / or with diabetic retinopathy;
- 3) Poor control of blood pressure in hypertensive patients (defined as blood pressure >150/95mmHg, including antihypertensive medication);

- 4) With surgical contraindication due to other local or systemic conditions at screening or baseline;
- 5) With any active ocular or periocular infection or inflammation (e.g., blepharitis, conjunctivitis, keratitis, scleritis, uveitis, endophthalmitis) at screening or baseline;
- 6) With uncontrolled glaucoma at screening or baseline (IOP  $\geq$  30mmHg when receiving medical treatment or as judged by the researchers);
- 7) With the presence of iris neovascularization or neovascular glaucoma at screening or baseline;
- 8) With ocular diseases which may interfere the study results at screening or baseline, including severe vitreous hemorrhage, peripheral retinal hole, proliferative diabetic retinopathy, proliferative vitreoretinopathy (≥ Level C), choroidal detachment;
- 9) With other causes which may result in macular hole associated-retinal detachment at screening or baseline, except high myopia;
- 10) Previously underwent scleral buckling surgery;
- 11) With current or planned medication known to have toxic effects on the lens, retina or optic nerve, including hydroxychloroquine, chloroquine, hydroxychloroquine, tamoxifen, phenothiazine and ethambutol;
- 12) With laboratory abnormalities, such as ALT, AST, TB, GGT, LDH, exceeded the normal limit by more than 2 times, and CREA or blood urea nitrogen exceeded 1.2 times the normal limit;
- 13) With abnormal coagulation function (defined as more than normal prothrombin time for 3 seconds or more, more than 1.5 of the international standard ratio (INR), activated partial thromboplastin time of 10 seconds or longer than the upper limit of normal time);
- 14) Patients who participated in any clinical study of medication within 3 months prior to screening (excluding vitamins and minerals)

### 6. Exit criteria

Exit criteria

- 1) Due to adverse events, especially severe adverse events, the researchers consider withdrawal of patients based on concerns of safety and ethics;
- 2) Drop out;
- 3) The patients voluntarily withdraw the informed consent;
- 4) Serious violation of the study protocol due to the subjects or investigators' reasons;
- 5) Other reasons that the researchers believe for quitting the study

### 7. Treatment

Group 1: The patients in Group 1 are treated by the surgical method of standard 3-port 23 gauge pars plana vitrectomy + internal limiting membrane peeling + air-fluid exchange + silicone oil infusion

Group 2: The patients in Group 2 are treated by the surgical method of standard 3-port 23 gauge pars plana vitrectomy + internal limiting membrane peeling + inverted internal limiting membrane insertion + air-fluid exchange.

## 8. Inspection and observation schedule

| Period | Screen ing period | Randomiz<br>ation<br>period | | Follow up period <sup>1</sup> | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseli | | V | V | V | V | V | V | V | Termina | Unsched |
| Project \ | ne | Treatment | 1 | 2 | 3 | 4 | 5 | 6 | 7 | tion | uled visit |
| Visiting | -7~0d | 0d | 1 | 1 | 2 | 4 | 8 | 12 | 6 | 12m | |
| time | -/~Va | va | d | w | w | w | w | w | m | 12111 | _ |
| Informed | × | | | | | | | | | | |
| consent | ^ | | | | | | | | | | |
| Inclusion | | | | | | | | | | | |
| and | × | × <sup>2</sup> | | | | | | | | | |
| exclusion | | ,, | | | | | | | | | |
| criteria | | | | | | | | | | | |

Version number: Version 2

| Demograp | | | | | | | | | | |
|-----------------|---|---|---|---|---|---|---|---|---|---|
| hic data | × | | | | | | | | | |
| Chief | | | | | | | | | | |
| complaint | | | | | | | | | | |
| and | × | | | | | | | | | |
| current | ^ | | | | | | | | | |
| medical | | | | | | | | | | |
| history | | | | | | | | | | |
| Medical | × | | | | | | | | | |
| history | ^ | | | | | | | | | |
| Previous | | | | | | | | | | |
| surgery/ | | | | | | | | | | |
| trauma | | | | | | | | | | |
| history | × | | | | | | | | | |
| and ocular | | | | | | | | | | |
| surgery | | | | | | | | | | |
| history | | | | | | | | | | |
| Diagnosis | × | | | | | | | | | |
| Vital signs | × | × | × | × | × | × | × | × | × | × |
| 3 | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ |
| General | | | | | | | | | | |
| physical | × | × | × | × | × | × | × | × | × | × |
| examinati | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ |
| on | | | | | | | | | | |
| Slit lamp | | | | | | | | | | |
| examinati | | | | | | | | | | |
| on <sup>4</sup> | × | | | | | | | | | |
| (binocular | | | | | | | | | | |
| ) | | | | | | | | | | |

| Slit lamp | | | | | | | | | | | |
|-----------------|---|---|---|---|---|---|---|---|---|---|---|
| examinati | | | | | | | | | | | |
| on <sup>5</sup> | | | × | × | × | × | × | × | × | × | × |
| (study | | | | | | | | | | | |
| eye) | | | | | | | | | | | |
| ECG and | | | | | | | | | | | |
| chest | × | | | | | | | | | | |
| radiograp | | | | | | | | | | | |
| hy <sup>6</sup> | | | | | | | | | | | |
| Laborator | | | | | | | | | | | |
| у | × | | | | | | | | | | |
| examinati | | | | | | | | | | | |
| on <sup>7</sup> | | | | | | | | | | | |
| Auxiliary | | | | | | | | | | | |
| examinati | × | | × | × | × | × | × | × | × | × | × |
| on <sup>8</sup> | | | | | | | | | | | |
| Low | | | | | | | | | | | |
| vision | | | | | | | | | | | |
| quality of | × | | | | | | × | × | × | × | |
| life | | | | | | | | | | | |
| questionn | | | | | | | | | | | |
| aire 9 | | | | | | | | | | | |
| History | | × | | | | | | | | | |
| change | | | | | | | | | | | |
| Randomiz | | × | | | | | | | | | |
| ation | | | | | | | | | | | |
| Surgical | | × | | | | | | | | | |
| treatment | | | | | | | | | | | |

| Subject | V | | | | | | | | | | |
|-------------|---|---|---|---|---|---|---|---|---|---|---|
| files | × | | | | | | | | | | |
| Adverse | | × | × | × | × | × | × | × | × | × | × |
| events 10 | | | ^ | ^ | ^ | ^ | ^ | ^ | ^ | | ^ |
| Previous / | | × | | | | | | | | | |
| combined | × | | × | × | × | × | × | × | × | × | × |
| medicatio | | | | | | | | | | | |
| n 11 | | | | | | | | | | | |
| Quit in | | | × | × | × | × | × | × | × | × | |
| advance | | | | | | | | | | | |
| Statistical | | | | | | | | | | | |
| summary | | | | | | | | | × | | |
| of major | | | | | | | | | | | |
| endpoints | | | | | | | | | | | |
| Summary | | | | | | | | | | | |
| of the | | | | | | | | | | × | |
| study | | | | | | | | | | | |
| Unschedul | | | | | | | | | | | × |
| ed visits | | | | | | | | | | | |
| Research | | | | | | | | | | | |
| statistics | | | | | | | | | | × | |
| summary | | | | | | | | | | | |

### Remarks

- (1) Visit Window: Visit 2 to visit 6; each visit has a window period of  $\pm 3$  days; visit 7 and end visit allow a window period of  $\pm 7$  days.
- (2) If both the eyes meet the requirements in the screening, the eye with the poorer BCVA should be selected as the study eye, unless for medical reasons, the researchers believe that the other eye is more suitable for the research.

  The study eye will undergo surgical treatment according to the protocol. If the BCVA damage of the contralateral eye is caused by macular hole associated with retinal detachment secondary to high myopia, according to the

judgment of the researchers, the contralateral eye can also be recommended for surgical treatment. The contralateral eye was labeled as the contralateral eye for treatment. The treatment of bilateral eyes should not be performed on the same day.

- (3) Vital signs, including blood pressure, pulse, respiration, armpit temperature, should be measured after sitting for 5 minutes.
- (4) Slit lamp examination: Use "Slit Lamp Examination Form-I" (Attachment 1). Accept the examination results carried out before the informed consent signature during the same hospitalization.
- (5) Slit lamp examination: Use "Slit Lamp Examination Form-II" (Attachment 2).
- (6) ECG, chest radiography: Accept the examination results carried out before the informed consent signature during the same hospitalization.
- (7) Laboratory examination includes routine blood test, blood biochemistry, routine blood coagulation, hepatitis B quantification, HCV antibody, TPPA+RPR and HIV antibody. Accept the examination results carried out before the informed consent signature during the same hospitalization.
- (a) Routine blood test: white blood cell, neutrophil, lymphocyte, neutrophil ratio, lymphocyte ratio, red blood cell, hemoglobin, platelet.
- (b) Blood biochemistry: alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, lactate dehydrogenase, gamma glutamyltransferase, total bilirubin, direct bilirubin, total protein, albumin, urea, creatinine, uric acid, glucose, triglyceride, total cholesterol, potassium, sodium, chloride, calcium, phosphorus.
- (c) Routine blood coagulation: prothrombin time, activated partial thromboplastin time, thrombin time, fibrinogen, prothrombin time -INR.
- (8) Auxiliary examinations:
- (a) Auxiliary examinations in the screening period include: BCVA OU, IOP OU, OCT of study eye, wide angle CP of study eye, the multifocal electroretinogram of study eye, microperimetry analysis of study eye, ocular axis measurement of study eye, B-scan ultrasound of study eye. Accept the examination results carried out before the informed consent signature during the same hospitalization.
- (b) Auxiliary examinations in V1 and 2 include: BCVA OU, IOP OU, OCT of study eye, wide angle CP of study ocular axial measurement of study eye;
- (c) Auxiliary examinations in V3 include: BCVA OU, IOP OU, OCT of study eye, wide angle CP of study eye, B-scan ultrasound of study eye;
- (d) Auxiliary examinations in V4 include: BCVA OU, IOP OU, OCT of study eye, wide angle CP of study eye;

(e) Auxiliary examinations in V5, 6, 7, end visits, and unscheduled visits include: BCVA OU, IOP OU, OCT of study eye, wide angle CP of study eye, the multifocal electroretinogram of study eye, microperimetry analysis of study eye and B-scan ultrasound of study eye.

(9) The low vision quality of life questionnaire: Subjects were asked to self-rate according to the low vision quality of life questionnaire (Attachment 3);

(10) Adverse events: Adverse events were collected from the time the subjects sign informed consent until the end of the study.

(11) Previous/ combined medication: Collect relevant information from the time the subjects sign informed consent until the end of the study, including all the medication used for the treatment of AE or SAE.

#### 9. Outcome Assessment

1) Primary Outcome Assessment:

Macular hole closure rate: Fundus examination combined with optical coherence tomography (OCT) are performed 3 months after surgery.

2) Secondary Outcome Assessment:

Best corrected visual acuity (LogMAR): 6 months after the surgery

Reattachment rate of retinal detachment: Use fundus examination combined with B-scan ultrasound, optical coherence tomography (OCT) to observe the reattachment rate of retinal detachment within 12 months after the surgery. (The reattachment rate assessment is performed 12 months after the first surgery among the patients with air tamponade. The reattachment rate assessment is performed 12 months after the first surgery among the patients with silicone oil tamponade, and the silicone oil removal is performed 6 months after the previous surgery.)

Postoperative complication rate

#### 10. Adverse event

(1) Adverse events (AE) refer to any adverse event that occurs during clinical studies, but do not necessarily have causal relationship with the surgery.

Safety evaluation should be carried out from the signature of the informed consent until the end of the study, according to management requirements (Adverse events or serious adverse events should be reported).

(2) Severe adverse events (SAE) refer to the occurrence of hospitalization, prolonged

hospitalization, disability, incapacity, life-threatening or death, congenital malformations during the clinical trials.

(3) Record of adverse events

During the study, all adverse events should be recorded. Records should include the name of AE (using the standard medical terminology), the date of AE occurrence and disappearance / stablization, severity, impact on the surgery, relationship with the surgery, treatment measures and outcomes.

(4) Reports of serious adverse events

If serious adverse events occur, researchers must fill in the report of serious adverse events. The report should be signed and dated, and be reported to the ethics committee within 24 hours.

### 11. Target case load and sample size calculation

Target case load: 38

The study uses the superiority design. According to the references and the professional judgment, macular hole closure rate is 25% in the control group (group 1), while in the experimental group (group 2), macular hole closure rate is 65%. The significant level  $\alpha$  is 0.05, and test performance (1- beta) is 0.80. The software of NCSS PASS 14 is used, and each group has 17 cases with the loss rate of 10%. The final sample size is 38.

#### 12. Randomization

Stratified randomization is conducted according to the extent of retinal detachment [type 1 (within the arcade area), type 2 (beyond the arcade area)]. The software of NCSS PASS 14 will be used. The study includes 2 groups.

### 13. Masking method

In this study, the third party independent evaluation method is used to evaluate the results of the study. The analyzer is in the masking state, and the patients and the surgeons are in the nonmasking state.

### 14. Statistical data processing

(1) Validity analysis: Descriptive statistical method is used to describe the research indicators. Univariate analysis of continuous variables is performed using ANOVA, and univariate analysis of categorical variables is performed using chi square test. The repeated measurement data are

analyzed by mixed effect model. The population of effectiveness analysis is the population of people with intention to be treated.

(2) Safety analysis: The safety assessment of clinical parameters (including adverse events, laboratory tests, vital signs, etc.) will be carried out. Descriptive statistics method is adopted. The

safety analysis of the population is the population of all groups received treatment.

(3) Subgroup analysis: To determine whether the therapeutic effects of different subgroups are

consistent, the component outcomes (and 95% confidence interval (CI)) are estimated for the major

endpoints within the subgroup of the following categorical variables:

The type of retinal detachment [type 1 (within the arcade area), type 2 (beyond the arcade area)]

Gender (male and female)

15. Study implementation period (Anticipated)

April 7<sup>th</sup>, 2017 to April 6<sup>th</sup>, 2020

16. Quality Control

The researcher and laboratory personnel involved in this project must have the professional

knowledge and experience required in the study protocol;

The researchers and other staff involved in the study perform their duties, and strictly follow the

clinical trial plan and adopt standard operating procedures to ensure the implementation of the

quality control and quality assurance system;

To ensure that the data is complete, accurate, authentic and reliable, all the relevant observation

results and findings need to be verified in each phase of the clinical trials;

The researchers and other staff who participated in the study have sufficient time and reliable

sources of subjects for the study;

For all examinations, examination room conditions must meet the requirements: clean, quiet,

and no pollution; Pipeline arranged neatly; Safety management measures, emergency and first-aid

facilities are all required; Instruments placed properly; Dustproof, shockproof, appropriate special

ventilation and exhaust facilities are required; For the instruments sensitive with the change of

temperature and humidity, there is a constant temperature and dehumidification device; The

examination room responsible personnel with corresponding professional theory and practical

experience, can effectively organize, guide and carry out business, and be responsible for the study results; Different inspection instruments are operated by specially-assigned staff, and regular verification is required.

The specimen involved in the study are collected by specially-assigned staff;

The procedure is checked according to the standard operating procedures;

When the study protocol needs to be modified, ethical committees should be convened according to standard operating procedures, and the functions of the ethics committee should be fully applied to ensure the interests of the subjects to be protected;

Set up data files and keep all the original data according to the requirements of the scheme in chronological order for verification;

The inspectors regularly check the related activities and documents, to evaluate whether the study is operated according to the study protocol, standard procedures and relevant laws and regulations, and whether the test data is recorded timely, truly, accurately and completely. The inspection should be carried out by personnel not involved in the study, and the audit report shall be written. Meetings should be held with relevant personnel to discuss the problems found in the audit.

Version number: Version 2

**Specific Study Protocol** 

Overall objective

To evaluate the surgical outcomes of inverted internal limiting membrane insertion combined

with air tamponade in the treatment of macular hole retinal detachment (MHRD) in high myopia,

and also to compare the treatment efficacy between different surgical approaches of MHRD.

Main study contents

This study uses a new surgical method (vitrectomy combined with inverted internal limiting

membrane insertion) to evaluate its effect on the prognosis of macular hole retinal detachment

secondary to high myopia.

This study uses a new surgical method (intraocular sterilized air tamponade) to assess its effect

on the prognosis of macular hole retinal detachment secondary to high myopia.

This study compares this new type of surgery with the current commonly used surgery

(vitrectomy combined with internal limiting membrane peeling + silicone oil infusion) on the

prognosis of macular hole retinal detachment secondary to high myopia.

Study protocol

Title:

A Single Center, Randomized and Controlled Clinical Study of Inverted Internal Limiting

Membrane Insertion Combined with Air Tamponade in the Treatment of Macular Hole Retinal

Detachment in High Myopia

Key word:

Surgical procedures, air tamponade, high myopia, macular hole retinal detachment

Study design:

Single center, randomized, controlled, interventional, prospective

Aim:

The aim of this study is to evaluate the effectiveness and safety of different surgical procedures for

patients with macular hole retinal detachment secondary to high myopia.

**Primary Outcome Measure:** 

To evaluate the effectiveness of different surgical procedures by evaluating the following

indicators:

Macular hole closure rate: Fundus examination combined with optical coherence tomography

(OCT) are performed 3 months after surgery.

**Secondary Outcome Measure:** 

To evaluate the effectiveness and safety of different surgical procedures by evaluating the

following indicators:

Best corrected visual acuity (LogMAR): 6 months after the surgery

Reattachment rate of retinal detachment: Use fundus examination combined with B-scan

ultrasound, optical coherence tomography (OCT) to observe the reattachment rate of retinal

detachment within 12 months after the operation.(The reattachment rate assessment is performed

12 months after the first surgery among the patients with air tamponade. The reattachment rate

assessment is performed 12 months after the first surgery among the patients with silicone oil

tamponade, and the silicone oil removal is performed 6 months after the previous surgery.)

Postoperative complication rate of ocular adverse events

Postoperative complication rate of the non ocular adverse events

Postoperative complication rate of severe adverse events

**Key inclusion criteria** 

Prior written consent is required before any assessment.

Study eye selection criteria:

Visual impairment is caused by macular hole associated with retinal detachment secondary to high myopia

Axial length  $\geq$  26mm, or the refractive error  $\geq$  -6.0D

**Key exclusion criteria** 

Exclusion criteria for general medical history:

Local or systemic surgical contraindications at screening or baseline

For both eyes:

With any ocular eye or periocular infection or inflammation (e.g., blepharitis, conjunctivitis,

keratitis, scleritis, uveitis, endophthalmitis) at screening or baseline;

With uncontrolled glaucoma at screening or baseline (IOP ≥ 30mmHg when receiving medical

treatment or as judged by the researchers);

With the presence of iris neovascularization or neovascular glaucoma at screening or baseline.

For research eye:

With ocular diseases which may interfere the study results at screening or baseline, including

severe vitreous hemorrhage, peripheral retinal hole, proliferative diabetic retinopathy, proliferative

vitreoretinopathy ( ≥ Level C ), choroidal detachment;

With other causes which may result in macular hole associated-retinal detachment at screening

or baseline, except high myopia;

Previously underwent scleral buckling surgery.

Exclusion criteria for past or current systemic drug use:

With current or planned medication known to have toxic effects on the lens, retina or optic nerve,

including hydroxychloroquine, chloroquine, hydroxychloroquine, tamoxifen, phenothiazine and

ethambutol.

Study design

This study is a prospective, randomized, controlled study, involving multiple visits within 12

months. The patients with macular hole retinal detachment secondary to high myopia are randomly

divided into 2 treatment groups:

Group 1: The patients in Group 1 are treated by the surgical method of standard 3-port 23 gauge

pars plana vitrectomy + internal limiting membrane peeling + air-fluid exchange + silicone oil

infusion

Group 2: The patients in Group 2 are treated by the surgical method of standard 3-port 23 gauge

pars plana vitrectomy + internal limiting membrane peeling + inverted internal limiting membrane

insertion + air-fluid exchange

Sample size calculation

The study uses the superiority design. According to the references and the professional

judgment, macular hole closure rate is 25% in the control group (group 1), while in the experimental

group (group 2), macular hole closure rate is 65%. The significant level ais 0.05, and test

performance (1- beta) is 0.80. The software of NCSS PASS 14 is used, and each group has 17 cases

with the loss rate of 10%. The final sample size is 38.

**Grouping method** 

Patients are assessed whether they meet the inclusion/exclusion criteria before inclusion. The

clinical research center completes the compliance assessment form, preoperative consents and

informed consent. Informed consent is a qualified standard, since it is agreed by the subjects to be

selected, randomly assigned, and agreed to complete the regular follow-up after the surgery.

1) Informed consent of the subjects

In this study, researchers must explain the research purpose, process, possible profit and risk

to the subjects (or the legal representative, or witnesses). Only when the subjects (or the legal

representative, or witnesses) fully understand the study, and sign informed consent, can they be

selected.

The informed consent form should be signed by the subjects (or their legal representatives or

witnesses) and the researcher who executed the informed consent procedure in two copies, each of

which has one copy.

2) Allocation of screening number of subjects

The subjects who signed the informed consent will be assigned to a screening number. The

center will assign a number of 4 Arabia numbers to each subject, with individual uniqueness. Among

them, the first number represents the clinical center number, and the second, third, fourth number is

the ordinal number, which is assigned to each subject according to the chronological order of the

informed consent agreement. The subjects name writing rules: When the name is consisted with two

characters, fill in the first two letters of each phonetic alphabet; When the name is consisted with

three characters, fill in the first letters of each phonetic alphabet and the second letter of the third

phonetic alphabet; When the name is consisted with four characters, fill in the first letters of each

phonetic alphabet; When the name is consisted with five or more than five characters, fill in the first

letters of the first four phonetic alphabets.

Randomized controlled clinical trial design is used in this study.

Randomization: Stratified randomization is conducted according to the type of retinal

detachment [type 1 (within the arcade area), type 2 (beyond the arcade area)]. The software of NCSS

PASS 14 will be used. The study includes 2 treatment groups.

According to randomization procedures, the researchers assign ID numbers to patients. The

ID number of the randomization group must be recorded together with the patient screening number

in a random directory. Completed random directory should be signed and hand over to the data

center by the researcher.

Masking method

In this study, the third party independent evaluation method is used to evaluate the results of

the study. The analyzer is in the masking state, and the subjects and the surgeons are in the non-

masking state.

**Outcome evaluation** 

1) Primary Outcome Measures:

To evaluate the effectiveness of different surgical procedures by evaluating the following

indicators:

The difference between macular hole closure rate, closed type in each group from baseline to

the 3rd month

2) Secondary Outcome Measures:

To evaluate the effectiveness and safety of different surgical procedures by evaluating the

following indicators:

The difference of the reattachment rate of retinal detachment between each group from baseline

to the 6th month

The difference of the reattachment rate of retinal detachment between each group from baseline

to the 12th month

The change of BCVA relative to baseline and the difference between groups from baseline to

the 6th month

The change of BCVA relative to baseline and the difference between groups from baseline to

the 12th month

The number of people whose BCVA result improves by more than 1 row, 2 rows and 3 rows

comparing to the baseline at a time.

The number of people whose BCVA result decreases by 3 rows comparing to the baseline at a

time

The difference of multifocal ERG results between each group from 1 week to the 6th month

after surgery

The difference of multifocal ERG results between each group from 1 week to the 12th month

after surgery

The change of microperimetry analysis results from 1 week to the 6th month after surgery

relative to baseline, and the difference between each group

The change of microperimetry analysis results from 1 week to the 12th month after surgery

relative to baseline, and the difference between each group

The change of the extent of foveal ellipsoid zone damage from baseline to the 6th month after

the surgery relative to baseline, and the difference between each group

The change of the external limiting membrane integrity of fovea from baseline to the 6th month

after the surgery relative to baseline, and the difference between each group

Version number: Version 2

The change of the extent of foveal ellipsoid zone damage from baseline to the 12th month after

the surgery relative to baseline, and the difference between each group

The change of the external limiting membrane integrity of fovea from baseline to the 12th

month after the surgery relative to baseline, and the difference between each group

Describe the number of retreatment and retreatment modalities for patients with different

surgical procedures over a period of 12 months

Evaluate the safety of different surgical procedures by assessing the type, frequency and

severity of ocular adverse events and non-ocular adverse events or severe adverse events during 12

months

Data analysis

(1) Validity analysis: Descriptive statistical method is used to describe the research indicators.

Univariate analysis of continuous variables is performed using ANOVA, and univariate analysis of

categorical variables is performed using chi square test. The repeated measurement data are

analyzed by mixed effect model. The population of effectiveness analysis is the population of people

with intention to be treated.

(2) Safety analysis: The safety assessment of clinical parameters (including adverse events,

laboratory tests, vital signs, etc.) will be carried out. Descriptive statistics method is adopted. The

safety analysis of the population is the population of all groups received treatment.

(3) Subgroup analysis: To determine whether the therapeutic effects of different subgroups are

consistent, the component outcomes (and 95% confidence interval (CI)) are estimated for the major

endpoints within the subgroup of the following categorical variables:

The type of retinal detachment [type 1 (within the arcade area), type 2 (beyond the arcade area)]

Gender (male and female)

**CRC** assistance

The study requires one to two clinical research coordinator (CRC)

Responsiblities:

(1) Contact the subjects before 3-7 days before a follow-up;

(2) Communicate with the director in advance, and make appointments for patient follow-ups;

(3) Arrange the relevant examination for the patients;

(4) Have good communication skills;

(5) Fill in Case Report Form.

Benefit status of subjects

The therapy in this study may help to further control the patient's condition, to optimize the

treatment of the disease, to provide the necessary advice for the future treatment of patients, to

provide useful information for treatment or disease;

If the subjects quit the study, the doctors will still perform the related examinations and

treatments to ensure the safety of the subjects.

**Risk supervision** 

The principal investigator and researchers should make full use of the informed consent when

asking the patient to participate in the clinical trial. They should confirm that the patients fully

understand its content, participate in this study based on the their free will, and sign the informed

consent. The principal investigator, researchers and participants should sign on the informed consent

form respectively.

During the implementation process of the clinical trials, if serious adverse events (including

the events such as the occurrence of hospitalization, prolonged hospitalization, disability, incapacity,

life-threatenning or death, congenital malformation during the process of the clinical trial) occur,

the events must be promptly reported to the center of clinical trials and the principal investigator.

When the subjects suffer any health impairment caused by the study, researchers undertake the

cost of treatment and the corresponding economic compensation for clinical trial-related injury or

death, except the impairment caused by medical accidents.

## Research schedule

| Time | Schedule |
|---|---|
| 2017.4~2018.3 | Enroll patients, observe patients, collect clinical data, complete |
| | international clinical trial registration (clinicaltrial.gov), and complete |
| | midterm summary of patients who completed the first year visit |
| 2018.4~2019.3 | Follow patients up and collect clinical data |
| 2019.4~2020.4 | Complete the visit of all patients, complete the analysis of clinical data, |
| | subject summary, and prepare acceptance. |

Version number: Version 2

## **Technology Roadmap**



## **Attachment 1**

## Slit Lamp Examination Form (right eye)-I

| Whether to have | Whether to have slit lamp examination (right eye)?: $_1\Box Yes \rightarrow Please$ record as follows, $_0\Box No$ |
|---|---|
| Other lesions of | ₀□No |
| eyelid | 1□Yes, Please describe: |
| 1. Conjunctiva (right eye) | |
| | <sub>0</sub> □Normal. It may appear white or reddish pink, without peripheral congestion. |
| | The conjunctival or bulbar conjunctival vessels are easily |
| | observed |
| | 1□Slight redness, reddish color, mainly confined to the palpebral conjunctiva |
| Congestion | or bulbar conjunctiva |
| Congestion | 2□Mild redness, reddish color, mainly confined to the conjunctiva or bulbar |
| | conjunctiva |
| | 3□Moderate, palpebral conjunctiva or bulbar conjunctiva is bright red |
| | 4□Severe, palpebral conjunctiva or bulbar conjunctiva is deep diffuse bright |
| | red |
| | <sub>0</sub> □Normal, no swelling |
| | 1□Slight, beyond normal and regional |
| Edema | 2□Mild, mild conjunctival swelling, beyond normal, regional |
| | 3□Moderate, conjunctival swelling moderately |
| | 4□Severe, large conjunctival swelling |
| | <sub>0</sub> □Nil, no bleeding |
| Subconjunctival | ¹□Slight, flat and less than 1 quadrant |
| Subconjunctival | 2□Mild, bulging, and 1 quadrant, or flat and more than 1 quadrants |
| hemorrhage | 3□Moderate, bulging and >1 quadrant, but less than 2 quadrants |
| | 4□Severe, bulging and more than 2 quadrants |

| Other conjunctival lesions | 0□No 1□Yes, Please describe: |
|---|---|
| 2. Cornea (right e | eye) |
| Edema | o□Nil, transparent and clear □□Slight, micro and local epithelial haze □□Mild, turbid vitreous appearance and may contain tiny droplets □□Moderate, turbid vitreous appearance with a large number of vacuoles □□Severe, bullous and / or stromal edema, localized or diffuse, with or without matrix streaks |
| Other corneal | o□No |
| lesions | <sub>1</sub> □Yes, Please describe: |

# Slit Lamp Examination Form (right eye)-I

| 3. Anterior chamber (right eye) | |
|---|---|
| | <sub>0</sub> □Nil, no cells |
| | <sub>1</sub> □Slight, 1-5 cells |
| Cell number | 2□Mild, 6-25 cells |
| | <sub>3</sub> □Moderate, 26-50 cells |
| | 4□Severe, the number of cells is too large to count |
| | <sub>0</sub> □Nil, no Tyndall effect |
| | 1□Slight, almost cannot distinguish the Tyndall effect |
| Anterior chamber flare | 2□Mild, slight brightness |
| | 3□Moderate, strong brightness |
| | 4□Severe, very strong and aqueous humor is white or milky |
| Other lesions | ₀□No |
| Other resions | 1□Yes, Please describe: |
| 4. Iris / pupil (right eye) | |
| Iris / pupil (right eye) | Clinically significant abnormality: 0 No 1 Yes, Please describe: |

| 5. Lens (right eye) | |
|---|---|
| | 1□Complete |
| Lens (right eye) | 2□Artificial |
| | <sub>3</sub> □Nil |
| Other lesions | ₀□No |
| Other lesions | 1□Yes, Please describe: |
| Transparency | |
| | ₀□Nil |
| | 1□There are turbidity, but below standard pictures |
| Cortex | 2□There are turbidity, and the severity of the standard picture is the |
| | same or more serious |
| | 3□Not applicable |
| | ₀□Nil |
| | 1□Turbid, but below standard pictures |
| Nucleus | 2 Turbid, the same or more serious than standard pictures |
| | 3□Not applicable |
| | <sub>0</sub> □Nil |
| | 1□Turbid, but below standard pictures |
| Posterior capsule | <sub>2</sub> Turbid, the same or more serious than standard pictures |
| | ₃□Not applicable |

## Slit Lamp Examination Form (right eye)-I

6. Vitreum (right eye)

| | <sub>0</sub> □Nil, no cells |
|---|---|
| | 1□Slight, 1-10 cells |
| Anterior vitreous cell | <sub>2</sub> □Mild, 11-30 cells |
| count | ₃□Moderate, 30-50 cells |
| | <sub>4□</sub> Severe, >50 cells |
| Othersheim | ₀□No |
| Other lesions | ¹□Yes, Please describe: |
| | ₀□Nil |
| Vitreous / anterior | ı□Slight |
| retinal hemorrhage | ₂□Mild |
| retinal nemormage | <sub>3</sub> □Moderate |
| | 4□Severe |
| 7. Macular and retina (right eye) | |
| | ₀□Nil |
| | <sub>1</sub> □Hole diameter≤1/3PD |
| Macular hole | <sub>2</sub> □Hole diameter>1/3PD, and≤1/2PD |
| | ₃□Hole diameter>1/2PD, and≤1PD |
| | 4□Hole diameter>1PD |
| | ₀□Nil |
| | <sub>1</sub> □Yes, Please describe: |
| Retinal detachment | <sub>1</sub> □Within the arcade |
| | 2□Beyond the arcade, and within the equator |
| | ₃□Beyond the equator |
| Peripheral retinal split | ₀□No |
| holes | 1□Yes, Please describe: |
| Posterior scleral | ₀□No |
| staphyloma | 1□Yes, Please describe: |
| Other lesions | ₀□No |
| | <sub>1</sub> □Yes, Please describe with words or pictures: |

| _ |
|---|

## **Attachment 1**

## Slit Lamp Examination Form (left eye)-I

| Whether to have slit lamp examination (left eye)?: ₁□Yes→Please record as follows, ₀□No | |
|---|---|
| Other lesions of | ₀□No |
| eyelid | ¹□Yes, Please describe: |
| 1. Conjunctiva (right eye) | |
| | <sub>0</sub> □Normal. It may appear white or reddish pink, without peripheral congestion. |
| | The conjunctival or bulbar conjunctival vessels are easily |
| | observed |
| | 1□Slight redness, reddish color, mainly confined to the palpebral conjunctiva |
| | or bulbar conjunctiva |
| Congestion | 2□Mild redness, reddish color, mainly confined to the conjunctiva or bulbar |
| | conjunctiva |
| | ₃□Moderate, palpebral conjunctiva or bulbar conjunctiva is bright red |
| | 4□Severe, palpebral conjunctiva or bulbar conjunctiva is deep diffuse bright |
| | red |
| | <sub>0</sub> □Normal, no swelling |
| | 1□Slight, beyond normal and regional |
| Edema | 2□Mild, mild conjunctival swelling, beyond normal, regional |
| | 3□Moderate, conjunctival swelling moderately |
| | 4□Severe, large conjunctival swelling |
| | ₀□Nil, no bleeding |
| Subconjunctival | 1□Slight, flat and less than 1 quadrant |
| hemorrhage | 2□Mild, bulging, and 1 quadrant, or flat and more than 1 quadrants |
| | 3□Moderate, bulging and >1 quadrant, but less than 2 quadrants |

| | 4□Severe, bulging and more than 2 quadrants |
|---|---|
| Other | ₀□No |
| conjunctival | |
| lesions | ¹□Yes, Please describe: |
| 2. Cornea (left ey | re) |
| | <sub>0</sub> □Nil, transparent and clear |
| | 1□Slight, micro and local epithelial haze |
| Г1 | 2□Mild, turbid vitreous appearance and may contain tiny droplets |
| Edema | 3□Moderate, turbid vitreous appearance with a large number of vacuoles |
| | 4□Severe, bullous and / or stromal edema, localized or diffuse, with or without |
| | matrix streaks |
| Other corneal | ₀□No |
| lesions | ¹□Yes, Please describe: |

## Slit Lamp Examination Form (left eye)-I

| 3. Anterior chamber (left eye) | |
|---|---|
| | <sub>0</sub> □Nil, no cells |
| | ¹□Slight, 1-5 cells |
| Cell number | <sub>2</sub> □Mild, 6-25 cells |
| | ₃□Moderate, 26-50 cells |
| | 4□Severe, the number of cells is too large to count |
| | ₀□Nil, no Tyndall effect |
| | <sub>1</sub> □Slight, almost cannot distinguish the Tyndall effect |
| Anterior chamber flare | 2□Mild, slight brightness |
| | 3□Moderate, strong brightness |
| | 4□Severe, very strong and aqueous humor is white or milky |
| Other lesions | ₀□No |
| | ¹□Yes, Please describe: |
| 4. Iris / pupil (left eye) | |

Version number: Version 2

| Iris / pupil (right eye) | Clinically significant abnormality: 0□No1□Yes, Please describe: |
|---|---|
| 5. Lens (left eye) | |
| | ¹□Complete |
| Lens (right eye) | 2□Artificial |
| | <sub>3</sub> □Nil |
| Other lesions | ₀□No |
| Other resions | 1□Yes, Please describe: |
| Transparency | |
| | ₀□Nil |
| | 1□There are turbidity, but below standard pictures |
| Cortex | 2□There are turbidity, and the severity of the standard picture is the |
| | same or more serious |
| | ₃□Not applicable |
| | ₀□Nil |
| | 1□Turbid, but below standard pictures |
| Nucleus | <sub>2</sub> Turbid, the same or more serious than standard pictures |
| | 3□Not applicable |
| | ₀□Nil |
| | 1□Turbid, but below standard pictures |
| Posterior capsule | 2□Turbid, the same or more serious than standard pictures |
| | <sub>3</sub> □Not applicable |

# Slit Lamp Examination Form (left eye)-I

| 6. Vitreum (left eye) | |
|---|---|
| Anterior vitreous cell | <sub>0</sub> □Nil, no cells |
| | 1□Slight, 1-10 cells |
| | <sub>2</sub> □Mild, 11-30 cells |
| count | ₃□Moderate, 30-50 cells |
| | 4□Severe, >50 cells |
| Otherstein | ₀□No |
| Other lesions | ¹□Yes, Please describe: |
| | ₀□Nil |
| Vitreous / anterior | ı□Slight |
| | 2□Mild |
| retinal hemorrhage | <sub>3</sub> □Moderate |
| | 4□Severe |
| 7. Macular and retina (let | ft eye) |
| | $_{0}\square \mathrm{Nil}$ |
| | <sub>1</sub> □Hole diameter≤1/3PD |
| Macular hole | <sub>2</sub> □Hole diameter>1/3PD, and≤1/2PD |
| | <sub>3</sub> □Hole diameter>1/2PD, and≤1PD |
| | 4□Hole diameter>1PD |
| | ₀□Nil |
| | <sub>1</sub> □Yes, Please describe: |
| Retinal detachment | <sub>1</sub> □Within the arcade |
| | 2□Beyond the arcade, and within the equator |
| | ₃□Beyond the equator |
| Peripheral retinal split | ₀□No |
| holes | ¹□Yes, Please describe: |
| Posterior scleral | ₀□No |
| staphyloma | ¹□Yes, Please describe: |

| | ₀□No | | | | | | |
|---|---|---|---|---|---|---|---|
| Other lesions | <sub>1</sub> □Yes, | Please | describe | with | words | or | pictures: |

## **Attachment 2**

## Slit Lamp Examination Form (study eye)-II

| Whether to have slit lamp examination (study eye)?: ₁□Yes→Please record as follows, ₀□No | |
|---|---|
| Other lesions of | ₀□No |
| eyelid | ¹□Yes, Please describe: |
| 1. Conjunctiva (study eye) | |
| | <sub>0</sub> □Normal. It may appear white or reddish pink, without peripheral congestion. |
| | The conjunctival or bulbar conjunctival vessels are easily |
| | observed |
| | <sup>1</sup> □Slight redness, reddish color, mainly confined to the palpebral conjunctiva |
| Congestion | or bulbar conjunctiva |
| Congestion | 2□Mild redness, reddish color, mainly confined to the conjunctiva or bulbar |
| | conjunctiva |
| | 3□Moderate, palpebral conjunctiva or bulbar conjunctiva is bright red |
| | 4□Severe, palpebral conjunctiva or bulbar conjunctiva is deep diffuse bright |
| | red |
| | <sub>0</sub> □Normal, no swelling |
| | 1□Slight, beyond normal and regional |
| Edema | 2□Mild, mild conjunctival swelling, beyond normal, regional |
| | 3□Moderate, conjunctival swelling moderately |
| | 4□Severe, large conjunctival swelling |
| G 1 ' ' ' 1 | <sub>0</sub> □Nil, no bleeding |
| Subconjunctival | 1□Slight, flat and less than 1 quadrant |
| hemorrhage | 2□Mild, bulging, and 1 quadrant, or flat and more than 1 quadrants |

| | 3□Moderate, bulging and >1 quadrant, but less than 2 quadrants |
|---|---|
| | 4□Severe, bulging and more than 2 quadrants |
| Other conjunctival lesions | 0□No 1□Yes, Please describe: |
| 2. Cornea (study | eye) |
| Edema | o□Nil, transparent and clear □Slight, micro and local epithelial haze □Mild, turbid vitreous appearance and may contain tiny droplets □Moderate, turbid vitreous appearance with a large number of vacuoles □Severe, bullous and / or stromal edema, localized or diffuse, with or without matrix streaks |
| Other corneal | ₀□No |
| lesions | ¹□Yes, Please describe: |

## Slit Lamp Examination Form (study eye)-II

| 3. Anterior chamber (study eye) | |
|---|---|
| | <sub>0</sub> □Nil, no cells |
| | <sub>1</sub> □Slight, 1-5 cells |
| Cell number | <sub>2</sub> □Mild, 6-25 cells |
| | <sub>3</sub> □Moderate, 26-50 cells |
| | 4□Severe, the number of cells is too large to count |
| | <sub>0</sub> □Nil, no Tyndall effect |
| | 1□Slight, almost cannot distinguish the Tyndall effect |
| Anterior chamber flare | 2□Mild, slight brightness |
| | 3□Moderate, strong brightness |
| | 4□Severe, very strong and aqueous humor is white or milky |
| Other lesions | ₀□No |
| Other resions | ¹□Yes, Please describe: |

| 4. Iris / pupil (study eye) | |
|---|---|
| Iris / pupil (study eye) | Clinically significant abnormality: 0□No1□Yes, Please describe: |
| 5. Lens (studyeye) | |
| | ¹□Complete |
| Lens (study eye) | 2□Artificial |
| | <sub>3□Nil</sub> |
| Other lesions | ₀□No |
| Other lesions | ¹□Yes, Please describe: |
| Transparency | |
| | ₀□Nil |
| Cortex | 1□There are turbidity, but below standard pictures 2□There are turbidity, and the severity of the standard picture is the same or more serious 3□Not applicable |
| Nucleus | o□Nil 1□Turbid, but below standard pictures 2□Turbid, the same or more serious than standard pictures 3□Not applicable |
| Posterior capsule | o□Nil 1□Turbid, but below standard pictures 2□Turbid, the same or more serious than standard pictures 3□Not applicable |

## Slit Lamp Examination (study eye)-II

| 6. Vitreum (study eye) | |
|---|---|
| Anterior vitreous cell | <sub>0</sub> □Nil, no cells |
| | 1□Slight, 1-10 cells |
| | <sub>2</sub> □Mild, 11-30 cells |
| count | ₃□Moderate, 30-50 cells |
| | 4□Severe, >50 cells |
| Other lesions | $_{0}\square \mathrm{No}$ |
| Other lesions | ¹□Yes, Please describe: |
| | $_{0}\square \mathrm{Nil}$ |
| Vitreous / anterior | ı□Slight |
| | <sub>2</sub> □Mild |
| retinal hemorrhage | <sub>3</sub> □Moderate |
| | 4□Severe |
| | ₀□Nil |
| | 1□≤30% |
| Air volume in vitreous | <sub>2</sub> □>30%, and≤50% |
| cavity | ₃□>50%, and≤70% |
| | <sub>4</sub> □>70% |
| | 5□Not applicable |
| | ₀□Nil |
| Silicone oil volume in | 1□>50%, and≤70% |
| vitreous cavity | 2□>70%, and≤90% |
| vitreous cavity | 3□>90% |
| | 4□Not applicable |
| 7. Macular and retina (research eye) | |
| | ₀□Nil |
| Macular hole | <sub>1</sub> □Hole diameter≤1/3PD |
| Widediai noic | <sub>2</sub> □Hole diameter>1/3PD, and≤1/2PD |
| | <sub>3□</sub> Hole diameter>1/2PD, and≤1PD |

| | 4□Hole diameter>1PD |
|---|---|
| | ₀□Nil |
| | <sub>1</sub> □Yes, Please describe: |
| Retinal detachment | <sub>1</sub> □Within the arcade |
| | 2□beyond the arcade, and within the equator |
| | ₃□Beyond the equator |
| Peripheral retinal split | ₀□No |
| holes | ¹□Yes, Please describe: |
| Posterior scleral | ₀□No |
| staphyloma | 1□Yes, Please describe: |
| | ₀□No |
| Other lesions | 1□Yes, Please describe with words or pictures: |

## **Attachment 3**

## Low vision quality of life questionnaire

5=Nil; 4-2=Moderate; 1=Severe; x=Unable to do.

How well do you know about your current vision? 5=Much, 1=Little

| 1. Because of your vision, in the following circumstances, do you feel difficult?. | |
|---|---|
| 1. Feel tired (for example, only after a short time using eyes) | □5 □4 □3 □2 □1□x □Others |
| 2. At home at night | □5 □4 □3 □2 □1□x □Others |
| 3. Look at things in the right amount of light | □5 □4 □3 □2 □1□x □Others |
| 4. Feel the light glare (such as car lamp or sun make you dazzle) | □5 □4 □3 □2 □1□x □Others |
| 5. Look at road signs | □5 □4 □3 □2 □1□x □Others |
| 6. Watch TV (or enjoy pictures) | □5 □4 □3 □2 □1□x □Others |
| 7. Look at moving objects (such as cars on the road) | □5 □4 □3 □2 □1□x □Others |
| 8. Determine the distance or depth of objects | □5 □4 □3 □2 □1□x □Others |
| 9. See the stairs or railings | □5 □4 □3 □2 □1□x □Others |
| 10. Walk outdoors (e.g., on an uneven sidewalk) | □5 □4 □3 □2 □1□x □Others |
| 11. Cross the street when there is vehicles | □5 □4 □3 □2 □1□x □Others |
| 12. Generally speaking | □5 □4 □3 □2 □1□x □Others |
| 2. Because of your vision, so you | |
| 1. Not satisfied with your current life | □5 □4 □3 □2 □1□x □Others |
| 2. Be upset about not being able to do some work | □5 □4 □3 □2 □1□x □Others |
| 3. Visiting relatives and friends is limited | □5 □4 □3 □2 □1□x □Others |
| 4How well do you know about your current vision | □5 □4 □3 □2 □1□x □Others |
| 3. If you use visual aids or glasses, if there are difficulties when doing the following things | |
| 1.Identify uppercase fonts | □5 □4 □3 □2 □1□x □Others |
| 2. Read newspaper articles and books | □5 □4 □3 □2 □1□x □Others |
| 3. Read labels (for example, on a bottle or kit) | □5 □4 □3 □2 □1□x □Others |
| 4. Reading letters | □5 □4 □3 □2 □1□x □Others |

| 5. Use some tools (such as sutures or scissors) | □5 □4 □3 □2 □1□x □Others |
|---|---|
| 4. If you use visual aids or glasses, if there are difficulties when doing the following things | |
| 1. Watch the clock to know the time | □5 □4 □3 □2 □1□x □Others |
| 2. Sign or write cards | □5 □4 □3 □2 □1□x □Others |
| 3. Identify your own handwriting | □5 □4 □3 □2 □1□x □Others |
| 4. Do daily activities (such as housework) | □5 □4 □3 □2 □1□x □Others |

## **Attachment 4**

## **Abbreviations**

| Abbreviations and special terms | Explanation |
|---|---|
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| BCVA | Best corrected visual acuity |
| CREA | Serum creatinine |
| Wide angle CP | Wide angle fundus color photography |
| GGT | Glutamyl transferase |
| HCV | Hepatitis C virus |
| HIV | Human immunodeficiency virus |
| LDH | Lactate dehydrogenase |
| LogMAR visual acuity | Standard logarithmic visual acuity |
| MHRD | Macular hole complicated with retinal detachment |
| INR | International normalized ratio |
| IOP | Intraocular pressure |
| OCT | Optical coherence tomography |

| OD | Right eye |
|----------|----------------------------------------------|
| OS | Left eye |
| OU | Both eyes |
| PDR | Proliferative diabetic retinopathy |
| PVR | Proliferative vitreoretinopathy |
| ТВ | Total bilirubin |
| TPPA+RPR | Treponema pallidum antibody gelatin particle |
| | agglutination test + syphilis serum test |
| VA | Vision acuity |